CLINICAL TRIAL: NCT04733677
Title: User Experience of the OSR M1 Reusable Elastomeric Air Purifying Respirator in Non-Clinical Settings
Brief Title: User Experience of the OSR M-1
Status: Terminated | Type: Observational
Why Stopped: NIOSH certification became impossible, so decision was made to terminate
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00070715
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: COVID; coronavirus; respirator; mask; N99
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OSR M-1 N95: All subjects will be fitted with an OSR M1 N95 mask

SUMMARY:
The purpose of this observational study is to verify the user acceptance of the Open Standard Respirator-Model 1 (OSR-M1) by clinicians through pre-trial survey and quantitative fit-testing and post-trial feedback surveys. This study will help to guide further design modifications and clarify quantities of employee populations that may benefit from elastomeric respirator use for the deployment of OSR M1 Air Purifying Respirators (APRs) in the Wake Health network.

DETAILED DESCRIPTION:
The study team hypothesizes that the OSR M-1 APR with National Institute for Occupational Safety and Health classification 99% Airborne Particle Filtration (N99) will have increased fit and seal as well as user comfort and acceptance over disposable National Institute for Occupational Safety and Health classification 95% Airborne Particle Filtration (N95) filter facepiece respirators (FFR). The study team is proposing to assess the acceptance and functional usability of the OSR-M1 in Wake Forest Baptist Health System as a N95 disposable FFR alternative for improved protection and economy.

1. Assess the effectiveness and causation of successful/unsuccessful fit testing of the OSR M1 APR by measuring anthropometry of facial features and performing quantitative fit testing of clinicians.
2. Determine usability, initial and long-term acceptance of the OSR M1 APR relative to standard issue disposable FFRs through user survey and assessment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical staff who are issued and routinely wear N95 FFR or equivalent APR's are eligible.

Exclusion Criteria:

* Participants unable to pass the fit testing will be excluded from the study.
* Anyone with a contraindication to wearing an N95 FFR (I.e. pregnancy, underlying medical conditions) will be excluded from the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Clinical staff who are issued and routinely wear N95 FFR may be screened.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Successful Fits | Day 1
  Percentage of subjects that pass fit-factor testing [0%-100%]
Quality of Fit Score | Day 1
  Scores can range from 0 to 10000 with a higher score denoting a better fit. A score of 100 qualifies as a successful OSHA half-mask respirator fit test.
Percentage of Participants that Fit in a Small Size Mask | Day 1
  percentage [0%-100%]
Percentage of Participants that fit in a Medium Size Mask | Day 1
  percentage [0%-100%]
Percentage of Participants that fit in a Large Size Mask | Day 1
  percentage [0%-100%]
User Acceptance Percentage | Day 10
  Percentage of participants that prefer the experimental device over currently used device [0-100%]

SECONDARY OUTCOMES:
Percentage of Impression Change | Baseline through Day 10
  Changes in impression of the device (pre-trial vs. post-trial) - percentage of positive or negative change [-100% - +100%]

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Brown, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No